CLINICAL TRIAL: NCT06982027
Title: Assessment of Peripheral Regional Anesthetic Blockade Using a Non-Invasive Surface Electromyogram (EMG) on the Affected and Unaffected Extremity
Brief Title: Peripheral Regional Blockade and EMG
Acronym: Electromyogram
Status: Enrolling by invitation | Phase: Not Applicable | Type: Interventional
Sponsor: Nationwide Children's Hospital (Other)
Responsible Party: Principal Investigator, Grant Heydinger, Principal Investigator - MD, Nationwide Children's Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: STUDY00004642
Record Dates: First submitted 2025-05-13; First posted 2025-05-21 (Actual); Last update posted 2025-10-30 (Actual); Status verified 2025-10

CONDITIONS: Surgery

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes

ARMS (1):
- General Anesthesia with peripheral regional block (Experimental): All patients will have general anesthesia and a peripheral regional block (upper or lower extremity block). EMG electrodes will be placed on both the extremity to be blocked in two dermatomes within the sensory distribution of the nerve and then in the same two sensory dermatomes on the contralateral extremity that is not being blocked.
  Interventions: Device: BlockSynop surface electromyography device; Procedure: Peripheral nerve block

INTERVENTIONS:
Device: BlockSynop surface electromyography device — The EMG monitor uses non-invasive surface electrodes that measures electrical activity in response to muscle stimulation. After all electrodes have been placed on the patient, the electrodes will be connected to a prototype non-significant risk device (NSR) BlockSynop surface electromyography device and monitoring of sEMG signal will begin. The device is a non-invasive and non-significant risk device.
Procedure: Peripheral nerve block — An injection of numbing medicine near a specific nerve or group of nerves to numb the part of the body undergoing surgery.

SUMMARY:
The investigators are studying a type of technology that is already used called surface electromyography (EMG). This measures and records electrical activity using sensor stickers in a non-invasive way. The purpose of this study is to use a prototype/test surface EMG machine to measure how well regional anesthesia (nerve block) is working. This device is non-invasive and being used for research use as an unapproved medical device. The information may teach us how to give nerve blocks more safely and effectively.

Study participation: Subjects having surgery will have the surface EMG sensor stickers placed on their arms or legs before surgery. These will stay on during surgery and for part of recovery.

Study visits: The study will consist of 1 visit that starts in the pre-operative area, through the surgery, and for part of recovery time after surgery.

DETAILED DESCRIPTION:
This study aims to investigate how non-invasive, non-significant risk EMG monitoring can be used intraoperatively to objectively characterize peripheral nerve blockade (upper or lower extremity) in pediatric, adolescent, and young adult patients undergoing surgery. We also aim to quantify the impact of sevoflurane (general anesthesia) on basal muscle tone based on EMG changes.

Hypothesis: EMG monitoring can be utilized to objectively measure neuraxial blockade, including onset, resolution, density, and dermatomal level.

ELIGIBILITY:
Inclusion Criteria:

* Patients ≤ 21 years of age
* Patient presenting for a surgical procedure in which GA and a peripheral regional block will be used

Exclusion Criteria:

* Patients > 21 years of age
* Parent / patient refusal
* Premature infants; neuromuscular disease; systemic infection; hemodynamic instability; coagulation disorder; degenerative CNS abnormality that precludes regional anesthesia; and local anesthetic allergy; pregnant women.

Ages: 0 Years to 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 100 (Estimated)
Dates: Start 2025-09-03 (Actual); Primary Completion 2027-01 (Estimated); Study Completion 2027-12 (Estimated)

PRIMARY OUTCOMES:
Determine onset of peripheral nerve blockade + general anesthesia using surface EMG as measured by power of signal amplitude. | Preoperative placement through resolution of motor blockade in the PACU. Timeframe being day of surgery- up to one day.
  Performance of non-invasive surface EMG following administration of peripheral nerve blockade + general anesthesia. This will be assessed by EMG signal amplitude.
Determine resolution of peripheral nerve blockade + general anesthesia using surface EMG as measured by power of signal amplitude. | Preoperative placement through resolution of motor blockade in the PACU. Timeframe being day of surgery - up to one day.
  Performance of non-invasive surface EMG following administration of peripheral nerve blockade and general anesthesia. This will be assessed by EMG signal amplitude.
Determine density of peripheral nerve blockade + general anesthesia using surface EMG as measured by power of signal amplitude. | Preoperative placement through resolution of motor blockade in the PACU. Timeframe being day of surgery - up to one day.
  Performance of non-invasive surface EMG following administration of peripheral nerve block and general anesthesia. This will be assessed by EMG signal amplitude.

SECONDARY OUTCOMES:
Quantify the impact of sevoflurane (%) on basal muscle tone based on EMG signal amplitudes. | Intraoperative time frame. Timeframe being day of surgery.
  Quantify the impact of sevoflurane (%) on basal muscle tone based on EMG signal amplitudes.

CONTACTS AND LOCATIONS:
Overall Officials: Grant Heydinger, MD, Principal Investigator — Nationwide Children's Hospital
Locations (1):
- Nationwide Children's Hospital, Columbus, Ohio, United States